CLINICAL TRIAL: NCT04607343
Title: Clinical Trial of a Rehabilitation Device Based on Electrical Stimulation for Patients With Obstructive Sleep Apnoea (OSA): a Study Protocol
Brief Title: Clinical Trial of a Rehabilitation Device Based on Electrostimulation for Obstructive Sleep Apnoea
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resourses
Sponsor: Fundación Neumologica Colombiana (Other)
Collaborators: Universidad de la Sabana (Other)
Responsible Party: Principal Investigator, Luis F. Giraldo-Cadavid, MD, PhD. Pulmonary Medicine, Interventional Pulmonology, Fundación Neumologica Colombiana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201803 23403
Record Dates: First submitted 2020-09-22; First posted 2020-10-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnoea
Keywords: Rehabilitation device; Electrical stimulation; Genioglossus muscle; Laryngopharyngeal sensory test
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Electrostimulation begins with electrodes placed on the skin in the submental and submandibular triangles, making sure not to place electrodes on the carotid sinus. The goal of this stimulation will be topographical closeness of the genioglossus, geniohyoid, mylohyoid, platysma and digastric muscles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental): Patients will undergo a conventional flexible nasopharyngeal laryngoscopy in which the degree of obstruction and the laryngopharyngeal sensitivity during wakefulness will be determined. Electrostimulation will be applied at different submandibular points with increasing intensity until the contraction of the dilation muscles of the airway or until the patient cannot tolerate the electrostimulation. The presence of contraction of stimulated muscles will be determined by external and endoscopic inspection.
  Interventions: Device: Rehabilitation device based on electrical stimulation

INTERVENTIONS:
Device: Rehabilitation device based on electrical stimulation — Experimental tests with transcutaneous electrical stimulation at different intensities and at the points of the submandibular region previously explored will be conducted first of all on the five healthy volunteer subjects. During these tests, the neuromuscular thresholds of the upper airway, the most effective points of electrostimulation and the tolerance of intervention will be determined. The determination of the functional threshold will be made by clinical evaluation of the subject during stimulation.

SUMMARY:
The aim of this study is to evaluate in a clinical trial a rehabilitation device for patients with obstructive sleep apnoea (OSA) based on oropharyngeal electrical stimulation, which strengthens the dilating muscles of the upper airway, improves mechanical laryngopharyngeal sensitivity and improves OSA. Furthermore, to perform experimental electrotherapy, nasoendoscopy, polygraphy and polysomnography tests with the device in order to calculate thresholds of functional and sensory intensities on the dilating muscles of the upper airway in patients with OSA. These tests also include the detection of signals that measure breathing events during sleep in patients with OSA in order to use them in the control mechanisms of the electrostimulation device. Assess the effects and safety of the device in a group of five healthy volunteers for preliminary results. Finally, to evaluate in a small group of patients with OSA the device capacity to stimulate the upper-airway dilating muscles and to reduce the Apnea-Hypopnea Index (AHI) and oxygen desaturation indices when the electrostimulation device is used over a medium-term period (eight weeks) with morning and evening therapy sessions.

DETAILED DESCRIPTION:
Obstructive sleep apnoea-hypopnoea syndrome (OSA) is a respiratory disorder characterised by repetitive obstruction of the upper airway, leading to several interruptions during sleep. It is currently one of the main public health problems worldwide and one of the main cardiovascular risk factors in developed and intermediate developing countries, whose populations are increasing in obesity and age.

One of the common treatments for OSA is continuous positive airway pressure (CPAP) devices, which pumps air through a hose, reaches a mask that the patient has over his or her nose and travels the airway, keeping the upper airway open during sleep and avoiding episodes of airway collapse. The problem is that CPAP is not accepted by some patients due to a lack of adaptation, so alternative treatments may be needed. For some years, there have been explorations of treatments related to electrical stimulation of the muscles of the upper airway as therapy to reduce the number of episodes of apnoea (measured through the apnoea-hypopnoea index) during the night, strengthening these muscles through stimulation.

This is the protocol of a clinical study of a rehabilitation device for home use that not only provides functional stimulation of the upper-airway dilator muscles but also provides sensory stimulation. This device works by strengthening the dilating muscles of the upper respiratory tract and improving the sensory capacity of the laryngo-pharyngeal tract and is based on existing publications on the effectiveness of functional and somatosensory neurostimulation through neuroplasticity in the recovery of neurological deficits.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with confirmed OSA (four with mild OSA, four with moderate OSA and four with severe OSA) who sign their informed consent to participate in the study.

Exclusion Criteria:

* Pregnancy
* Basal polysomnography that does not meet validity criteria to be interpreted.
* Anticoagulation (although not a contraindication for laryngopharyngeal sensory endoscopic testing, anticoagulation is an exclusion criterion for this study to maintain the lowest level of risk).
* Haemorrhagic diathesis (to avoid risk of severe epistaxis during nasal endoscopy).
* Glasgow scale less than 15 (to avoid confusion with sensory or motor laryngopharyngeal involvement due to neurological disease that compromises the state of consciousness).
* Basal oxygen saturation by awake pulse oximetry below 88%.
* Patients with more than 5% of the total apnoea events being of central origin. (to avoid including patients with central sleep apnoea in whom laryngopharyngeal electrostimulation would have no effect).
* Inflammatory or infectious lesions on the face or neck
* Skin hypersensitivity
* Anaesthetic areas, burns, bruises or recent wounds in the area of electrical stimulation
* Cardiac pacemakers or other telemetry-controlled devices,
* History of maxillofacial or pharyngeal surgery.
* Active cancer
* Tumours of the laryngopharyngeal tract.
* Significant mental and/or behavioural conditions or inability of the patient to cooperate during the examination/intervention.
* Epilepsy
* Central Nervous System (CNS) surgery in the last three months (to avoid confusion with muscle or sensory laryngopharyngeal compromise).
* Brain trauma in the last three months (to avoid confusion with muscle or sensory laryngopharyngeal compromise).
* Neurological sequelae of any cause compromising the head and neck muscles (to avoid confusion with muscle or sensory laryngopharyngeal compromise).
* Underlying neuromuscular diseases affecting the head and neck muscles (to avoid confusion with muscle or sensory laryngopharyngeal involvement due to neuromuscular disease).
* Chronic use of systemic corticosteroids at doses greater than or equal to 20 mg daily of prednisone or equivalent (to avoid confusion with corticosteroid myopathy that compromises the laryngopharyngeal region).
* Bone prostheses or osteosynthesis (in polarized currents there is danger of chemical burn and bone resorption)
* Acute febrile processes
* Chronic decompensated diseases
* Diseases in terminal states
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of the apnoea-hypopnea index (AHI) during sleep | 2 months
  A median reduction of 10 on the AHI is expected with the intervention.

SECONDARY OUTCOMES:
Desaturation index | 2 months
  number of desaturations per hour during sleep.
sleep time spent under 90% oxygen saturation (T90) | 2 months
  Percentage of sleep time spent under 90% oxygen saturation.
oxygen saturation by pulse oximetry (SpO2) nadir | 2 months
  Lowest oxygen saturation by pulse oximetry.
Mean SpO2 | 2 months
  Mean oxygen saturation by pulse oximetry.
Number of patients who lower one or more categories in the severity of OSA | 2 months
  Moving from severe to moderate, severe to mild or moderate to mild OSA or normalising the AHI
Number of patients who climb one or more categories in the severity of OSA | 2 months
  Moving from mild to moderate, mild to severe or moderate to severe OSA
Improvement in the Sleep Apnoea Quality of Life Index (SAQLI) | 2 months
  Improvement in the quality of life as measured by the SAQLI
Improvement in the Epworth Sleepiness Scale (ESS) | 2 months
  Improvement in daytime sleepiness as measured by the ESS

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Giraldo, MD, PhD, Study Director — Fundación Neumológica Colombiana
Locations (2):
- Colombia (2):
  - Fundacion Neumologica Colombiana, Bogotá, Bogota D.C.
  - Universidad de La Sabana, Chía, Cundinamarca

IPD SHARING:
Plan to Share IPD: No
The patients clinical data will be entered into an anonymized database hosted on RedCap platform

REFERENCES:
- [Background] Caples SM, Gami AS, Somers VK. Obstructive sleep apnea. Ann Intern Med. 2005 Feb 1;142(3):187-97. doi: 10.7326/0003-4819-142-3-200502010-00010. No abstract available. PMID 15684207
- [Background] Gallas S, Marie JP, Leroi AM, Verin E. Sensory transcutaneous electrical stimulation improves post-stroke dysphagic patients. Dysphagia. 2010 Dec;25(4):291-7. doi: 10.1007/s00455-009-9259-3. Epub 2009 Oct 24. PMID 19856025
- [Background] Gillick BT, Zirpel L. Neuroplasticity: an appreciation from synapse to system. Arch Phys Med Rehabil. 2012 Oct;93(10):1846-55. doi: 10.1016/j.apmr.2012.04.026. Epub 2012 May 18. PMID 22613094
- [Background] Guilleminault C, Hill MW, Simmons FB, Dement WC. Obstructive sleep apnea: electromyographic and fiberoptic studies. Exp Neurol. 1978 Oct;62(1):48-67. doi: 10.1016/0014-4886(78)90040-7. No abstract available. PMID 729676
- [Background] Howlett OA, Lannin NA, Ada L, McKinstry C. Functional electrical stimulation improves activity after stroke: a systematic review with meta-analysis. Arch Phys Med Rehabil. 2015 May;96(5):934-43. doi: 10.1016/j.apmr.2015.01.013. Epub 2015 Jan 26. PMID 25634620
- [Background] Kezirian EJ, Boudewyns A, Eisele DW, Schwartz AR, Smith PL, Van de Heyning PH, De Backer WA. Electrical stimulation of the hypoglossal nerve in the treatment of obstructive sleep apnea. Sleep Med Rev. 2010 Oct;14(5):299-305. doi: 10.1016/j.smrv.2009.10.009. Epub 2010 Jan 29. PMID 20116305
- [Background] Schulte W, Scholze H, Werries E. Specificity of a cysteine proteinase of Entamoeba histolytica towards the alpha 1-CB2 peptide of bovine collagen type I. Mol Biochem Parasitol. 1987 Aug;25(1):39-43. doi: 10.1016/0166-6851(87)90016-8. PMID 2890103
- [Background] Page SJ, Cunningham DA, Plow E, Blazak B. It takes two: noninvasive brain stimulation combined with neurorehabilitation. Arch Phys Med Rehabil. 2015 Apr;96(4 Suppl):S89-93. doi: 10.1016/j.apmr.2014.09.019. PMID 25813373